CLINICAL TRIAL: NCT04136613
Title: Immediate Post Placental Insertion of Intrauterine Device at Cesarean Delivery, is Acceptable, Feasible and Safe in Iraqi Women.
Brief Title: Utility of Immediate Post Placental Insertion of Intrauterine Device During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taghreed Alhaidari (Other)
Collaborators: Elweyia Maternity Teaching Hospital (Other)
Responsible Party: Sponsor-Investigator, Taghreed Alhaidari, Assistant Professor/ Consultant Obstatricain & Gynecologist / Head of Scientific Affairs Unit, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9 Al-KindyCM
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Contraception Behavior
Keywords: Long acting reversible contraception; Post placental insertion of intrauterine device; Cesearean section; Safety; Feasibility
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post placental intra uterine device insertion (Experimental): There was immediate post-partum insertion of CuT 380 A intrauterine device after delivery of placenta during cesarean delivery. To overcome the considerable expulsion rate in the previous studies, we stabilize the IUD in place at the fundus be an absorbable suture; vicryl 0 that was introduced through the fundus, held the needle with sponge holder that was introduce up the fundus and taken out the vicryl through the lower uterine inscion, cutting the needle, hold the vicryl around the the T arm of the IUD and withdrawn back to be placed inside the fundus. Before closing the uterine incision, the threads were placed in the lower uterine segment, then the uterine incision was then closed routinely.
  Interventions: Device: Copper Intra uterine contarceptive device ( Cu-T 380A)

INTERVENTIONS:
Device: Copper Intra uterine contarceptive device ( Cu-T 380A) — Insertion of the Cu-T 380A during cesarean delivery immediately after placental removal.

SUMMARY:
Iraq is a country that ranks 33rd around world population growth rate. Meanwhile it is one of the counties in the middle east with the highest fertility rate, In addition to the considerable number of unintended pregnancy mainly in postpartum period.

The less use of family planning methods, the higher the fertility rate and the less interpregnancy interval which will carry an obvious more risk to the mother and the fetus especially if the cesarean delivery rate shown an increase trend as the case in Iraq. For that reason, contraception needs to be practiced in this critical period and an intrauterine contraceptive device ( IUD), the most commonly used reversible method of contraception worldwide could be an excellent choice during this period.

There were few evidences available about the safety and feasibility on practicing this type of contraception when we did start three years ago and no previous evidences in Iraq about practicing this method at the immediate postpartum period.

DETAILED DESCRIPTION:
Setting and design:

It is a single arm prospective clinical trial. That had been conducted at Al Elweyia Maternity Teaching Hospital and Al Hayat Private Hospital in Baghdad during the period from Sept., 1st, 2015 to Jan.,1st, 2019. Women delivering in those hospitals fulfilling inclusion criteria were included in the study after obtaining informed consent. The study protocol was approved by the ethical committee.

Data collection:

180 women were enrolled in the study, only 150 of them completed the study as thirty women we couldn't reach them through their contact numbers.

Intervention:

They had immediate post-partum insertion of Copper IUD (Cu-T 380A) after delivery of placenta immediately at cesarean delivery. To overcome the considerable expulsion rate in the previous studies, we stabilize the IUD in place at the uterine fundus by an absorbable suture; vicryl 0 that was introduced through the fundus ( from out to in), held the needle with sponge holder that was introduce up the fundus and taken out the vicryl through the lower uterine incision, cutting the needle, warped the vicryl around the the T arm of the IUD and withdrawn back to be placed inside the uterine cavity near the fundus. Before closing the uterine incision, the threads were placed in the lower uterine segment, then the uterine incision was closed routinely.

Follow up:

Women were assessed before discharge from the hospital looking for any excessive bleeding and were provided with a mobile number to call, in case she has any problem with the device that had been inserted.

Women were reassessed at six weeks postpartum, where speculum examination was done and if IUD threads was seen, they were trimmed at 2 cm from external os, otherwise if the threads of IUD were not seen a pelvic ultrasonography was done to confirm the presence of IUD in situ.

Women then were reassessed at yearly intervals for 3 years, looking for the occurrence of excessive bleeding during subsequent menstruation, for abdominal pain and abnormal vaginal discharge, missed threads, expulsion rate, continuation rate and how far they do recommend this method of contraception for other women.

Statistical analysis:

The data analyzed using Statistical Package for Social Sciences (SPSS) version 25. The data presented as mean, standard deviation and ranges. Categorical data presented by frequencies and percentages. Chi square test was used to assess the association between complication of IUD and certain information. Significance level was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivered by caesarean section whether elective or emergency, counseled for IUD insertion in pre- natal period or at the time of labour and who has the will and her husband to be engaged in the study.

Exclusion Criteria:

* Women with positive test for STIs (e.g. gonorrhea or chlamydia) in this pregnancy.
* Uterine anomaly that was known to distort the uterine cavity; whether uterine fibroid or congenital uterine anomalies.
* Developed postpartum hemorrhage.
* Diagnosed chorioamnionitis, intrapartum fever, or ruptured membranes for greater than 24 hours prior to delivery.
* Placenta previa or accrete.
* Anemia during pregnancy (Hb < 10 g/dl).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Number of the women accept to be engaged in this services. | First 6 months of the study
  Assessing the acceptability of the women for the service of IUD insertion during the immediate postpartum period after cesarean delivery.
Cost of IUD insertion during the immediate postpartum period. | Up to 3 years.
  Assessing the cost for the insertion of the device in the immediate postpartum period.
Time spent for IUD insertion during the immediate postpartum period | Up to 3 years
  Assessing the extra time spent for the insertion of the device in the immediate postpartum period.

SECONDARY OUTCOMES:
Percentage of Immediate complications | First 48 hours post cesarean section.
  Number of the women having immediate complications including excessive blood loss before discharge from the hospital.
Percentage of other complications | Six months and yearly up to 3 years
  Number of the women having heavy menstrual blood loss, abdominal pain, abnormal vaginal discharge, missed threads, perforation and expulsion rate.

CONTACTS AND LOCATIONS:
Overall Officials: Taghreed K Alhaidari, CABOG, Study Chair — Al Kindy College of Medicine, University of Baghdad; Taghreed K Alhaidari, CABOG, Principal Investigator — Al Kindy College of Medicine, University of Baghdad; Asmaa T Majeed, FICOG, Principal Investigator — Al Kindy College of Medicine, University of Baghdad; Sahar J Al-Jassani, CABOG, Principal Investigator — Al Kindy College of Medicine, University of Baghdad; Hayder A Fawzi, FICMS, Principal Investigator — Department of Pharmacy, Al-Esraa University College
Locations (1):
- Al Kindy College of Medicine/ University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No